CLINICAL TRIAL: NCT06936254
Title: One-Year Effect on Levodopa Equivalent Daily Dose of Thalamic VIM Nucleus Stimulation Compared to Subthalamic Nucleus Stimulation in Patients With Parkinson's Disease
Acronym: VIM vs NST
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, JARDEL Amory, Hospital Practitione, Central Hospital, Nancy, France
Other Study IDs: 2024PI211
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease (PD); Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VIM group: Patients in this group underwent deep brain stimulation (DBS) targeting the ventral intermediate nucleus (VIM) of the thalamus. VIM stimulation is primarily used for the control of tremor in Parkinson's disease patients, particularly those with tremor-dominant symptoms. This group includes individuals who were selected for DBS due to the prominence of tremor in their clinical presentation, with less emphasis on other motor symptoms such as bradykinesia or rigidity
- NST group: Patients in this group underwent DBS targeting the subthalamic nucleus (STN). STN stimulation is commonly used in patients with advanced Parkinson's disease, particularly for those who experience motor fluctuations, dyskinesias, and who require a significant reduction in dopaminergic medication. This group includes patients who were selected for DBS based on their overall motor symptoms, including bradykinesia and rigidity, with or without tremor predominance

SUMMARY:
This study compares the effects of deep brain stimulation (DBS) of the thalamic VIM nucleus versus the subthalamic nucleus (STN) on the levodopa equivalent daily dose (LEDD) in patients with Parkinson's disease. The goal is to determine whether VIM stimulation, typically used for tremor, can also reduce medication needs. It hypothesizes that STN stimulation leads to greater LEDD reduction, but VIM may offer moderate benefits in selected case

DETAILED DESCRIPTION:
Thesis Summary:

Deep brain stimulation (DBS) is a well-established therapeutic option for patients with advanced Parkinson's disease. The two most commonly targeted structures are the subthalamic nucleus (STN) and the ventral intermediate nucleus (VIM) of the thalamus. While STN stimulation is known to allow a significant reduction in the levodopa equivalent daily dose (LEDD), the effects of VIM stimulation on medication dosage remain less clear, particularly in patients selected for predominant tremor.

Objectives:

To compare the evolution of LEDD one year after DBS targeting the VIM versus the STN in patients with Parkinson's disease.

To assess whether VIM stimulation also enables a meaningful reduction in dopaminergic medication.

To contribute to refining surgical indications based on the patient's clinical profile.

Hypotheses:

STN stimulation leads to a greater reduction in LEDD compared to VIM stimulation.

VIM stimulation, though primarily used for tremor control, may result in moderate LEDD reduction in specific patient profiles.

Surgical target selection should be personalized, considering not only motor symptom control but also the impact on medication requirements.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* Underwent surgery for subthalamic nucleus (STN) or ventral intermediate nucleus (VIM) deep brain stimulation
* Surgery performed at CHRU of Nancy
* Surgery performed between 2014 (DxCare implementation) and 2024

Exclusion Criteria:

* No clinical diagnosis of Parkinson's disease
* No initial dopaminergic treatment
* Surgery not performed at CHRU of Nancy
* Death within 1 year following surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients with Parkinson's disease who underwent deep brain stimulation (DBS) surgery targeting either the subthalamic nucleus (STN) or the ventral intermediate nucleus (VIM) of the thalamus at the CHRU of Nancy between 2014 (DxCare arrivals) and 2024. Eligible patients must have a diagnosis of Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the levodopa equivalent daily dose (LEDD) between Parkinson's disease patients undergoing deep brain stimulation (DBS) targeting the VIM thalamic nucleus versus the STN. | The primary endpoint, which is the change in levodopa equivalent daily dose (LEDD), will be measured one year post-surgery in both the VIM and STN DBS groups.
  To compare the one-year change in the levodopa equivalent daily dose (LEDD) between Parkinson's disease patients undergoing deep brain stimulation (DBS) targeting the VIM thalamic nucleus versus the STN.

CONTACTS AND LOCATIONS:
Locations (1):
- Chru Nancy, Nancy, Lorraine, France